CLINICAL TRIAL: NCT05338996
Title: Addressing Health Disparities in Engagement, Retention, and Utilization of PrEP Among South Florida Women of Color
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: Care 4 U Management, Inc. (Unknown); Care Resource Community Health Centers, Inc. (Unknown); Monarch Health Services, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-21-0499
Record Dates: First submitted 2022-03-07; First posted 2022-04-21 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: HIV Prevention; PrEP Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iENGAGE for PrEP (Experimental): We will conduct an exploratory pilot of the PrEP intervention, using a quasi-experimental design, among 80 multi-ethnic WOC in Miami-Dade, Broward, and Palm Beach counties to evaluate feasibility, acceptability, and fidelity. PrEP uptake, adherence, and retention in care will be measured over a 4-month period, including biomarkers of adherence.
  Interventions: Behavioral: iENGAGE for PrEP

INTERVENTIONS:
Behavioral: iENGAGE for PrEP — This intervention originally developed for people living with HIV (PLWH), is designed to promote engagement, retention, and adherence to treatment by addressing the social determinants of health that often act as barrier to remaining in care and achieving viral suppression. Based on our experience with this intervention we believe that it is well suited to similarly promote engagement, retention, and utilization of PrEP care among our proposed target population of WOC by a) removing barriers to care and b) addressing unmet needs by providing c) point-to-point linkage to care services delivered by multi-disciplinary teams of individuals within or outside of the health facility, and d) the use of telehealth visits to facilitate engagement in care and improve health visit attendance. The original iENGAGE is a 4-session, in-clinic behavioral intervention.

SUMMARY:
Women of color (WOC) in South Florida, the region with the highest HIV rates in the U.S., experience significant barriers to accessibility, uptake, and utilization of Pre-exposure prophylaxis (PrEP) for HIV prevention, despite FDA approval since 2012. The purpose of this study is to use a Community-Based Participatory Research (CBPR) approach to finalize, and pilot-test a multi-component evidence-based intervention to reduce health disparities in engagement, utilization, and retention in PrEP care, with the goal of improving HIV prevention outcomes for the target population of WOC in S. Florida, primarily African American, Latina, and Haitian women in 3 designated Ending the HIV Epidemic (EHE) counties: Miami-Dade, Broward, and Palm Beach counties.

DETAILED DESCRIPTION:
The purpose of this study is to use a Community-Based Participatory Research (CBPR) approach to finalize, and pilot-test a multi-component evidence-based intervention to reduce health disparities in engagement, utilization, and retention in PrEP care, with the goal of improving HIV prevention outcomes for the target population of WOC in S. Florida. We will conduct an exploratory pilot of the PrEP intervention, using a quasi-experimental design, among 80 multi-ethnic WOC in Miami-Dade, Broward, and Palm Beach counties to evaluate feasibility, acceptability, and fidelity. PrEP uptake, adherence, and retention in care will be measured over a 4-month period, including biomarkers of adherence. Adult women initiating or returning to PrEP services at our collaborating sites will be recruited, consented, enrolled and complete baseline assessments. They will participate in an adapted Integrating ENGagement and Adherence Upon Entry (iENGAGE) intervention to address social determinants of health barriers to maintaining PrEP care.

ELIGIBILITY:
Inclusion Criteria:

1. >=18 years of age;
2. female and identifying as female gender;
3. able to provide informed consent;
4. willing to document a negative HIV antibody test before starting PrEP;
5. reporting recent sexual risk (e.g., sex without condoms in last 3 months, sexually transmitted infection (STI) diagnosis in the last 6 months, post-exposure prophylaxis (PEP) use in the last 12 months, transactional sex, partners who are HIV+);
6. report history of alcohol and other drug (AOD) use in last 3 months;
7. willing to screen for medical contraindications to PrEP according to Florida Health Department guidelines;
8. currently not cognitively impaired;
9. reporting no history of bipolar disorder, psychosis, or current need for inpatient psychiatric hospitalization.

Exclusion Criteria:

1. Less than 18 years of age;
2. not female at birth
3. unable to provide informed consent;
4. unwilling to document a negative HIV antibody test before starting PrEP;
5. unwilling to screen for medical contraindications to PrEP according to Florida Health Department guidelines;
6. currently cognitively impaired;
7. reporting recent history of bipolar disorder, psychosis, or inpatient psychiatric hospitalization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female at birth and identifying as female gender
Enrollment: 72 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Percentage of women | Baseline
  We will measure the percentage of women who, having been invited for screening, complete the screening and enroll in the study.
Monthly Change in self-reported PrEP Adherence from Baseline to 4 month follow up | Monthly through study completion, an average of 4 months
  In measuring adherence, we will use a self-report questionnaire to assess the of number of missed doses in the last 7 days assessed at baseline, at each monthly intervention session and at the 4 month follow-up.
Monthly Change in concentration of Tenofovir measured by urine biomarker | Monthly through study completion, an average of 4 months
  In measuring adherence, we will also use point of care urine testing to evaluate short-term Tenofovir concentration (for those prescribed Tenofovir) at each monthly visit to compare with self-report data.
Concentration of Tenofovir measured by dried blood spot test | 4 month follow up
  In measuring adherence, we will also use dried blood spot testing for longer-term Tenofovir levels (for those prescribed Tenofovir) at the 4-month follow up assessment.
Percentage of participants retained in PrEP Care | 4 month follow up from those enrolled in the study.
  Retention in PrEP Care will be considered the percentage of women who complete the 4-month follow up assessment from those who enrolled in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jessy G Dévieux, PHD, Principal Investigator — Florida International Univ.
Locations (3):
- United States (3):
  - Care 4 U Community Health Center, Miami, Florida
  - Care Resource, Inc., Miami, Florida
  - Monarch Health Services, Inc., West Palm Beach, Florida

IPD SHARING:
Plan to Share IPD: Yes
In accordance with NIH guidelines, a data set will be created that cab be obtained by other investigators that does not include participants' identifying information. Investigators whose proposed use of the data has been approved by their institution's IRB will be allowed to request the dataset.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: When the primary data analysis of the study is finished.
Access Criteria: Institutional Review Board (IRB) approval; commitment to using data only for research purposes; commitment to securing the data using appropriate computer technology; commitment to destroying or returning the data when analyses are completed.